CLINICAL TRIAL: NCT06342271
Title: Effects of a Nordic Walking Program on Arm Swing Asymmetry and Temporospatial Gait Parameters Compared to Free Walking in People With Parkinson's Disease
Brief Title: Effects of Nordic Walking and Free Walking on Arm Swing Parameters and Gait in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Responsible Party: Principal Investigator, Jéssica Espinoza Araneda, Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-2023
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Arms swing; Gait; Gait Disorders, Neurologic; Nordic Walking; Rehabilitation
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Walking group (Experimental): The group will be training with a Nordic Walking protocol for 12- weeks, two times a week, completing 24 one-hour sessions.
  Interventions: Other: Nordic walking training
- Free Walking group (Active Comparator): The group will be training with a Free Walking protocol for 12- weeks, two times a week, completing 24 one-hour sessions.
  Interventions: Other: Free Walking training

INTERVENTIONS:
Other: Nordic walking training — Participants will receive Nordic walking training (to walk with poles) for 12 weeks, 3x/week.
  Arms: Nordic Walking group
Other: Free Walking training — Participants will receive Free walking training (to walk without poles) for 12 weeks, 3x/week.
  Arms: Free Walking group

SUMMARY:
People with Parkinson's Disease(PD) present a series of alterations such as muscle stiffness and motor slowing, which gradually affect the swinging movement of the arms and legs, altering the ability to walk, increasing the risk of falling, and reducing functionality. This implies a higher energy cost and a greater probability of developing freezing of the gait.

Nordic walking (NW) is a form of physical exercise characterized by the use of walking poles, which could contribute positively to arm swing movement and, thus, gait.

This clinical trial aims to compare Nordic Walking with free walking (FW) protocol training and investigate their effects on arm swing and gait parameters in people with PD.

The study hypothesizes that NW training will reduce asymmetry and increase arm swing amplitudes during gait to a greater extent than FW. Also, improvements in arm swing could positively influence lower limb performance during regular gait, increasing gait speed, stride length, functional mobility, and quality of life.

People with PD will complete 24 supervised NW or FW training sessions for 12 weeks. Both trainings will be identical in volume and intensity, the only difference will be the use of poles in the NW group. Blinded researchers will conduct evaluations at baseline (T0), post-intervention (T1), and in one-month follow-up (T2).

DETAILED DESCRIPTION:
Primary aims: To compare the effects of Nordic Walking (NW) with a free walking (FW) protocol training on arm swing in people with Parkinson's disease.

Secondary aims: To compare the effects of NW and FW protocol training on the performance of lower limbs during walking, functional mobility, and quality of life in people with Parkinson's disease.

Methodology Study design: randomized controlled clinical trial, parallel, single-blinded. The participants will be invited through posters disseminating the research. Each interested person will be contacted by telephone and invited to the Human Movement Sciences Laboratory of the University of Talca. After signing informed consent, the baseline evaluations will be carried out. A brief questionnaire containing bio-demographic information and health history will be completed to verify the inclusion and exclusion criteria. To establish the disease's stage, the Hoehn and Yahr scale will be applied. The cognitive status will be assessed with the Montreal Cognitive Assessment (MoCA).

After the baseline evaluation, a number will be assigned a number to each participant, and performed a randomization process into blocks of four participants to assign them to study groups.

Twenty-eight people with PD, stages 1-3 on the Hoehn and Yahr scale, will be randomly assigned to the NW training (n = 14) or FW training group (n = 14), according to a sample size calculation, with a 1:1 allocation ratio, matched by disease stage (stages I, II, and III). The distribution will be blinded to the evaluators and statisticians.

Interventions:

The training will be developed on the athletics track and trails of the University of Talca, Chile. The participants will be trained in groups (NW or FW), for 12 weeks, two times a week on alternate days, completing 24 one-hour sessions. The protocol will be standardized for both groups.

Two physiotherapists, blinded to the study groups, will conduct the evaluations at T0 (baseline assessment), T1 (after 12 weeks of intervention), and T2 (one-month follow-up).

To characterize the sample, we will collect bio-demographic information and health data. To evaluate the progression of motor and non-motor symptoms in PD, the Movement Disorder Society (MDS)-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) will be applied. To safeguard the safety of the participants and prescribe the training individually, vital parameters will be assessed. The anthropometric profile will be established through weight, height, and body mass index. The upper and lower limbs' lengths are also measured (m). To assess walking speed, a 10-meter walk test will be applied, and to assess aerobic capacity, a 6-minute walk test will be carried out.

Two accelerometers placed at the wrist level will acquire the arm swing parameters. Arm swing is defined as a rotational movement of the arm, occurring during walking, and running in bipeds in opposite directions (anterior and posterior). With a validated AS algorithm, the amplitude of the arm swing for both upper limbs will be calculated. The arm swing asymmetry will be determined according to the symmetry index, considering the phases of oscillation detected in both arms simultaneously with an equation. The gait temporal-spatial parameters (gait speed and step length) will be acquired under the same test conditions and simultaneously to obtain the arm swing parameters, using a wireless sensor model G-walk® (BTS, Italy). Functional mobility will be measured through the timed up-and-go test (TUG). The quality of life will be assessed through the Parkinson's Disease Questionnaire (PDQ39).

Adherence will be monitored by recording attendance at training sessions. Fully adherent participants will be considered those who attend more than 80% of sessions. Adverse events will be monitored in each session and reported in the results.

Statistic analysis: Descriptive data analysis will be calculated for all variables in both groups at baseline (T0). The normality distribution will be verified. To investigate differences in arm swing parameters, a repeated measures analysis of variance will be performed. To determine intra- and intergroup differences, a Bonferroni post-hoc test will be applied. To estimate the relationship between kinematic parameters and the asymmetry of arm swing with lower limb parameters, Pearson's correlation coefficient will be used. Subsequently, a multiple regression analysis will be performed. In the case of a non-normal distribution, non-parametric tests will be used. For the treatment of missing data, an imputation method using regression will be used. All results with a p-value lower than 0.05 will be considered statistically significant. Additionally, the size of the effect will be determined by Cohen's test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD, confirmed by a neurologist following the criteria of the Parkinson disease Society Brain Bank Criteria
* Age between 50-80 years
* Disease stage between I and III according to Hoehn and Yahr (Hoehn and Yahr)
* To be able to walk without technical aids.

Exclusion Criteria:

* Cognitive impairment (score < 26 in the Montreal Cognitive Assessment MoCA).
* Surgery lasting less than three months or deep brain stimulation (DBS).
* Presence of comorbidities that contraindicate moderate to high-intensity physical exercise.
* Participate in any walking training two or more times per week.
* Diagnosis of any other neurological or musculoskeletal condition that can cause motor compromise and interfere with locomotion.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the amplitude of arm swing | Before, after 12-weeks of training, and after one-month of follow-up.
  It is the movement of the arms in the antero-posterior direction during walking. Measurements will be made through accelerometers, and the unit of measurement will be degrees.
Change in the arm swing asymmetry | Before, after 12-weeks of training, and after one-month of follow-up.
  Asymmetry of the amplitude of movement between left and right swings during walking (0% means no asymmetry) [%]

SECONDARY OUTCOMES:
Change in the temporospatial measurements during walking including measurements of Gait speed [m/s] and step length [m]. | Before, after 12-weeks of training, and after one-month of follow-up.
  will be assessed using wireless IMU sensor model G-walk (BTS, Italy)
Change in the functional mobility will be measured through the Timed up and go (TUG). | Before, after 12-weeks of training, and after one-month of follow-up.
  TUG measures the function of the lower limbs, mobility, and risk of falling. It consists of a measurement of the time taken to complete a circuit of three meters in seconds.
Change in the quality of life | Before, after 12-weeks and after one-month of follow-up.
  Quality of life will be assessed through the Parkinson's Disease Questionnaire (PDQ39)

CONTACTS AND LOCATIONS:
Overall Officials: Jéssica Espinoza, PT, MsC, PhD, Principal Investigator — University of Talca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espinoza-Araneda J, Caparros-Manosalva C, da Cunha M, Marzuca-Nassr GN, Fritz-Silva N, Pagnussat AS. Nordic walking and arm swing asymmetry in people with Parkinson's disease: protocol for a randomised clinical trial. BMJ Open Sport Exerc Med. 2024 May 27;10(2):e002029. doi: 10.1136/bmjsem-2024-002029. eCollection 2024. PMID 38808265